CLINICAL TRIAL: NCT02657876
Title: An Open-Label, Prospective, Safety, and Tolerability Study of ExpressGraft-C9T1 Skin Tissue in the Treatment of Diabetic Foot Ulcers
Brief Title: ExpressGraft-C9T1 Skin Tissue as a Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C9T12015; R44DK069924-08 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2016-01-18 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Diabetes; Diabetic Foot Ulcer; Non-healing Wound
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ExpressGraft-C9T1 Skin Tissue (Experimental): Enrolled participants receive one application of ExpressGraft-C9T1 skin tissue
  Interventions: Biological: ExpressGraft-C9T1 Skin Tissue

INTERVENTIONS:
Biological: ExpressGraft-C9T1 Skin Tissue — ExpressGraft-C9T1 skin tissue is provided as a suturable, biologically-active, circular skin tissue with a fully-stratified epithelial compartment comprised of human keratinocytes (NIKSC9T1) and a dermal compartment containing fibroblasts

SUMMARY:
This study is designed as a prospective, open-label trial focused on assessing the safety and tolerability of ExpressGraft-C9T1 skin tissue in the treatment of diabetic foot ulcers (DFU). Because the focus is on safety rather than efficacy, a standard of care comparator is not included in this first-in-human study. Targeted enrollment for this study is up to 6 subjects with a confirmed diagnosis of diabetes and who have foot ulcers. Subjects will each receive a single application of ExpressGraft-C9T1 skin tissue on a single identified study DFU following a 10-14 day run-in period. Any subjects requiring additional treatment will receive protocol-defined dressings through Study Treatment Week 12 as necessary. Enrollment will occur with a minimum of one week between each subject.

ELIGIBILITY:
SUBJECT-SPECIFIC CRITERIA

1. Men and women 18 - 80 years of age, inclusive
2. Female subjects of childbearing potential must agree to practice birth control for the duration of the study
3. Documented Type 1 or Type 2 Diabetes Mellitus
4. HgbA1C ≤ 10.0%
5. Ankle:brachial blood pressure index (ABI) of 0.7 to 1.3

   * If ABI is > 1.3 (i.e., non-compressible ankle vessels) or cannot be measured, then Toe brachial index (TBI) of ≥ 0.5, or
   * Doppler arterial waveforms that are triphasic or biphasic at the ankle of affected leg
   * If ABI and TBI cannot be measured, then Transcutaneous pressure (TcpO2) of ≥ 40 around ulcer site, or
   * Skin perfusion pressure > 30 if neither ABI, TBI, nor TcpO2 can be measured near ulcer
6. Stable medications for 2 weeks prior to Study Treatment Day 0

   * Sliding scale insulin permitted
   * Select antimicrobial therapies can be used as needed
7. Capable and willing to attend the scheduled visits and comply with study procedures
8. Signed informed consent form (ICF) for study enrollment

   WOUND-SPECIFIC CRITERIA
9. Full-thickness ulcer on the foot of 1.0 cm^2 - 5.0 cm^2 at Screening Visit after debridement with no clinical signs and symptoms of infection. Full thickness is defined as penetrating the dermis, but not extending beyond the subcutaneous tissue.
10. Study ulcer has been present for at least 4 weeks but not more than 1 year

Exclusion criteria:

MEDICAL HISTORY/CURRENT MEDICAL CONDITION

1. Pregnant or nursing women
2. Prisoners
3. Abnormal laboratory value(s) for routine blood work that the Clinical Investigator deems would not be in the subject's best interest to participate
4. Osteomyelitis in the study ulcer foot in the last 30 days
5. Grade 3 or 4 lower extremity edema
6. Unable to tolerate off-loading
7. Active Charcot's foot
8. History of malignancy in previous 5 years, except for basal cell carcinoma that has been treated with local excision and is no longer present
9. Patients with unstable chronic renal disease or requiring dialysis
10. Gangrene in any part of study ulcer foot
11. Patients with a history of above- or below-knee amputation in the contralateral leg related to underlying chronic disease.

    * History of toe amputation in either leg would not be exclusionary.
12. Patients with history of poor compliance
13. Patients with baseline panel reactive antibody (PRA) of ≥ 20%

    MEDICATIONS/THERAPIES
14. Oral or parenteral corticosteroids, immunosuppressants, radiation therapy or chemotherapy within 30 days prior to study enrollment
15. Use of an investigational product within the preceding 60 days

    STUDY ULCER
16. Signs and symptoms of clinical infection at study ulcer site
17. Study ulcer requiring antimicrobial therapy at Screening Visit or Study Treatment Day 0 due to clinical suspicion of infection
18. Treatment of study ulcer with Regranex® or hyperbaric oxygen within preceding 30 days
19. Previous treatment of study ulcer with any cell and/or tissue product (CTP) therapy
20. Change in wound size (increase/decrease) greater than 25% from Screening Visit to Study Treatment Day 0
21. Other ulcers within 3 cm of study ulcer
22. Ulcers with tendon, muscle, joint capsule, or bone exposure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events through study completion | Through study completion, at approximately 12 months
  Clinically significant vital signs, infection, blood chemistry, hematology and immunological evaluations are recorded as adverse events during the study. The safety of ExpressGraft-C9T1 skin tissue will be evaluated by adverse events through the 12 month study session.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (1):
- SerenaGroup Research Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No